CLINICAL TRIAL: NCT06904274
Title: A Multi-center, Open Label, Randomized Parallel Group Study Evaluating the Proportion of Women With Complete Resolution of Nonatypical Endometrial Hyperplasia Treated With Mirena or Oral Medroxyprogesterone Acetate for 6 Months
Brief Title: Mirena for the Treatment of Nonatypical Endometrial Hyperplasia for 6 Months
Acronym: SUNFLOWER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22923
Record Dates: First submitted 2025-03-21; First posted 2025-04-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levonorgestrel (BAY865028, Mirena) (Experimental): Mirena will be inserted into the participant's uterus by the investigator on Day 1. At visit 4 (after 6 months) or if a participant discontinues her study participation prematurely, the Mirena will be removed by the investigator.
  Interventions: Combination Product: BAY865028
- Oral progestin (Active Comparator): Participants will receive 10mg oral progestin once daily, preferably always at the same time of the day, until visit 4 (after 6 months).
  Interventions: Drug: Medroxyprogesterone acetate

INTERVENTIONS:
Combination Product: BAY865028 — Intrauterine delivery system
  Arms: Levonorgestrel (BAY865028, Mirena)
Drug: Medroxyprogesterone acetate — Oral tablet
  Arms: Oral progestin

SUMMARY:
Researchers are looking for a better way to treat women with nonatypical endometrial hyperplasia (NAEH).

Endometrial hyperplasia is a condition where the lining of the uterus (called the endometrium) becomes too thick. Nonatypical means that the condition is not cancerous. It is often caused by hormone imbalances in women. Symptoms can include abnormal vaginal bleeding or irregular periods. If this condition is not treated, then it may lead to cancer.

Currently, there are no approved treatments for NAEH and that is why there is still an unmet medical need.

The study treatment, Mirena (also known as BAY 865028), is already available as a type of birth control device. It is inserted into the uterus where it gradually releases progesterone.

In this study, researchers want to find out if Mirena works for women with NAEH. They believe it can help by keeping hormone levels balanced in the body.

The main purpose of this study is to show that uterine lining goes back to completely normal lining after treatment with Mirena and that its use is safe in this population.

For this, the researchers will compare the number of participants with benign endometrium after 6 months of treatment with Mirena or oral MPA.

The study participants will be randomly assigned into one of two treatment groups. The randomization will be done 2:1 ratio, meaning that for every two participants assigned to Mirena, one will be assigned to oral medroxyprogesterone acetate (MPA). Based on their group, participants will receive Mirena, which is inserted into the uterus at the start of the study, or they will take progestins once daily by mouth for 6 months.

Each participant will be in the study for around 10 months with up to 5 visits to the study clinic/site.

Participants will visit the study clinic:

* once before the treatment starts
* 3 times with a gap of 3 months between the visits during the treatment
* then 1 more time after the treatment ends

During the study, the doctors and their study team will:

* check participant's health by performing tests such as blood and urine tests
* perform vaginal ultrasound and hysteroscopy. Hysteroscopy is a minor surgical procedure where a thin camera will be inserted into the womb to check for any abnormality. Sampling of the endometrial lining (cells in the womb) will be done with a thin tube at the same time.
* take samples of womb (endometrial) lining
* ask the participants questions about how they are feeling and what adverse events they are having

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Post-menarchal women (≥18 years) at the time of signing the informed consent.
* Women with histologically confirmed NAEH independent of their parity or menopausal status.

Exclusion Criteria:

* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results.
* Congenital or acquired uterine or cervical anomaly including fibroids, or cervical stenosis that in the opinion of the investigator, would interfere with insertion and/or retention of the intrauterine system (i.e., if they distort the uterine cavity).
* Use of any long-acting injectable sex-hormone preparations within 6 months prior to the start of study intervention, and /or short acting hormonal medication within 6 weeks prior to the start of study intervention.
* Pregnancy
* Participants with either known family or personal history of genetic predisposition to uterine, ovarian or colorectal cancers (e.g. Lynch syndrome).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population will be nulliparous and parous women (≥18 years of age) independent of their menopausal status.
Enrollment: 207 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2027-05-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Complete Resolution (CR) of NAEH | At 6 months
  Complete Resolution will be evaluated as benign endometrium.

SECONDARY OUTCOMES:
Recurrence of NAEH after CR | At 3 months follow up after 6 months treatment
  Recurrence of NAEH on 3 months treatment free after CR at 6 months
Progression after CR | At 3 months follow up after 6 months treatment
  Endometrial hyperplasia with atypia or endometrial cancer after 3 months treatment free follow up after CR at 6 months
Proportion of participants having hysterectomy | During treatment and 3 months follow up
Diagnosis of "benign endometrium" | At 6 months of treatment followed by 3 month treatment-free follow up
Number of participants with adverse events | From the signing of the informed consent form (ICF) up to 3 months after the last dose of study intervention
  All AEs will be coded using the latest version prior to database lock of the Medical Dictionary for Regulatory Activities

CONTACTS AND LOCATIONS:
Locations (80):
- United States (62):
  - UAB Medicine Center for Research in Women's Health, Birmingham, Alabama
  - Women's Health Alliance of Mobile, Mobile, Alabama
  - AMR - Mobile, AL, Mobile, Alabama
  - Velocity Clinical Research - Mobile, Mobile, Alabama
  - North Valley Women's Care, Glendale, Arizona
  - Mesa Obstetricians and Gynecologists | Research Department, Mesa, Arizona
  - Marchand OB/GYN, Mesa, Arizona
  - Velocity Clinical Research - Phoenix, Phoenix, Arizona
  - Cornerstone Clinic for Women - Aldersgate, Little Rock, Arkansas
  - Velvet Clinical Research, Burbank, California
  - Allen Clinical Research LLC, Gardena, California
  - UC Davis Health Lawrence J Ellison Ambulatory Care Center - OB/GYN, Sacramento, California
  - Alliance Clinical West Hills, West Hills, California
  - OB/GYN Department_Comprehensive Women's Health Center, Denver, Colorado
  - AMR - Fort Myers, FL, Fort Myers, Florida
  - Sweet Hope Research Specialty, Inc. - Hialeah, Hialeah, Florida
  - UF Health Women's Specialists - Emerson, Jacksonville, Florida
  - K2 Medical Research - South Orlando, Orlando, Florida
  - Entrust Clinical Research, Palmetto Bay, Florida
  - Emerald Coast Clinical Research, Panama City, Florida
  - Physician Care Clinical Research LLC | Sarasota, FL, Sarasota, Florida
  - USF Health South Tampa Center for Advanced Healthcare - Gynecology, Tampa, Florida
  - Paramount Research Solutions | College Park Location, Atlanta, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Women's Wellness / SKYCRNG, Chicago, Illinois
  - Office of Dr. Cindy Basinski, LLC, Newburgh, Indiana
  - McFarland Clinic - Medical Arts Building - OBGYN, Ames, Iowa
  - Velocity Clinical Research - Lafayette, Lafayette, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Gynecologic Oncology Associates, Shreveport, Louisiana
  - Omni Fertility and Laser Institute, Shreveport, Louisiana
  - Johns Hopkins Outpatient Center - Obstetrics and Gynecology, Baltimore, Maryland
  - Revive Research Institute - Michigan - Women's Health, Dearborn Heights, Michigan
  - Hutzel Women's Hospital, Detroit, Michigan
  - St. Dominic's Gynecology/Oncology, Jackson, Mississippi
  - SKY integrative Medical Center, Ridgeland, Mississippi
  - McGill Family Practice, Papillion, Nebraska
  - Affiliated Clinical Research, Inc. | Las Vegas, NV, Las Vegas, Nevada
  - Rutgers Robert Wood Johnson Medical School - OBGYN, New Brunswick, New Jersey
  - Bosque Women's Care | Albuquerque, NM, Albuquerque, New Mexico
  - Columbia University Medical Center - Gynecology, New York, New York
  - Montefiore Medical Park - Eastchester - OBGYN, The Bronx, New York
  - Reply OBGYN and Fertility PLLC, Durham, North Carolina
  - Unified Women's Clinical Research - Centre OB/GYN, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Axia Women's Health - Anderson Township, Cincinnati, Ohio
  - ClinOhio Research Services, LLC. | Columbus, OH, Columbus, Ohio
  - University Hospitals | UH Cleveland Medical Center - MacDonald Clinical Trials Unit, Mayfield Heights, Ohio
  - Bethesda North Hospital - Gynecology, Montgomery, Ohio
  - OB/GYN Associates of Erie, Erie, Pennsylvania
  - Chattanooga Medical Research, LLC. | Chattanooga, TN, Chattanooga, Tennessee
  - Paramount Research Solutions-Nashville, Nashville, Tennessee
  - South Texas Clinical Research, Corpus Christi, Texas
  - Discovery Clinical Trials - Dallas, Dallas, Texas
  - Progressive Women's Health Pllc, Friendswood, Texas
  - Biopharma Informatic - West Houston, Houston, Texas
  - UTHealth Womens Research Program | Memorial City, Houston, Texas
  - AIH Research- Broadway, Pearland, Texas
  - UVA Health Midlife Health and Gynecologic Specialties Northridge, Charlottesville, Virginia
  - Inova Fairfax Hospital - OBGYN, Falls Church, Virginia
  - Virginia Women's Health Associates, Reston, Virginia
- Canada (3):
  - The Ottawa Hospital, Riverside Campus - Department of Obstetrics, Gynecology and Newborn Care, Ottawa, Ontario
  - Sinai Health System - Obstetrics & Gynaecology, General Obs Gyn, Toronto, Ontario
  - Centres Investigation Clinique Mauricie, Trois-Rivières, Quebec
- China (15):
  - Chongqing Maternal and Child Health Care Hospital, Chongqing, Chongqing Municipality
  - Xiamen Maternity and Child Health Care Hospital - Gynecology Department, Xiamen, Fujian
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Women and Children's Hospital, Qingdao University - Gynecology department, Qingdao, Shandong
  - Chengdu Women & Children's Central Hospital, Chengdu, Sichuan
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital CAMS, Beijing
  - Foshan Women and Child Health Care Hospital, Foshan
  - The Third Affiliated Hospital of Southern Medical University - Gynecology Department, Guangzhou
  - Nanjing Medical University (NMU) - The Second Affiliated Hospital, Nanjing
  - Tangshan Maternal and Child Health Care Hospital, Tangshan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22923